CLINICAL TRIAL: NCT01988441
Title: The Influence of Autophagy on Nonalcoholic Fatty Liver Disease
Brief Title: The Influence of Autophagy on Fatty Liver
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 102066-F
Record Dates: First submitted 2013-11-07; First posted 2013-11-20 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Non-alcoholic Fatty Liver Disease; Obesity
Keywords: autophagy; children; polymorphism
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — serum, WBC DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is one of the most common causes of chronic liver disease worldwide. It is not known why only some obese subjects develop NAFLD. In recent years, a growing body of evidence showed a crucial role of autophagy in in the regulation of liver fat storage. The purpose of this study is to determine whether autophagy pathway-related genetic polymorphisms affect NAFLD.

DETAILED DESCRIPTION:
The investigators will perform a prospective comparison of the genotype distribution of autophagy pathway-related genetic polymorphisms between those with and without NAFLD in a cohort of obese children and adolescents.

[Subjects] Obesity is defined as the BMI value > 95 percentile by different age- and gender groups according to the standards of the Department of Health in Taiwan.

[Data collection] The following data were obtained for each subject: age, gender, BMI, waist and hip circumference. The investigators will measure total serum bilirubin, alanine aminotransferase, aspartate aminotransferase, γ-glutamyltransferase fasting glucose, triglyceride, total cholesterol, and high-density lipoprotein cholesterol, insulin, glucose, and adiponectin.

[Liver ultrasonography] All participants will receive an ultrasonographic study of the liver. NAFLD is defined as the presence of an ultrasonographic pattern consistent with the following criteria: liver-kidney echo discrepancy, attenuated echo penetration and visibility of diaphragm, and obscure hepatic vessel structures.

[Genotyping] Genomic DNA will be extracted from 3 cc venous blood from each participant. After extraction, the genomic DNA will be immediately stored at -80°C. The TaqMan genotyping assays will be performed for selected SNPs genotyping on ABI 7300 Real-Time PCR System (Applied Biosystems).

[Sample size] Sample size was estimated by Epi InfoTM 7 (CDC, USA) program. Because there was no previous data regarding to the effect of autophagy related gene on NAFLD, the investigators estimate the odds ratio to vary between 60-80%. The investigators used a confidence level of 95%, power of 80%, the ratio of controls to NAFLD cases of 25%, percent of controls exposed of 25-35%, the samples size required would be a total of 291-872 subjects.

ELIGIBILITY:
Inclusion criteria:

* Age 6-18 years old
* Obesity definition: BMI > 95% according to the age- and gender-specific standard by National Health Institute in Taiwan
* Willing to give written informed consent

Exclusion criteria:

* Alcohol consumption
* Chronic liver diseases, including hepatitis B, hepatitis C, Wilson disease and autoimmune hepatitis
* Major systemic diseases, including cardiopulmonary disease, renal failure, cancer, and psychotic disorder

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Obese Taiwanese children and adolescents
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2013-09; Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
The genotype distribution of autophagy pathway-related genetic polymorphisms between those with and without NAFLD | One year
  The genotype distribution of autophagy pathway-related genetic polymorphisms between those with and without NAFLD

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Cheng Lin, M.D., Ph.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided